CLINICAL TRIAL: NCT06113523
Title: Genetic Research of Monogenic Obesity in a Pediatric Cohort With Severe and Early Onset Obesity (GENOBE)
Acronym: GENOBE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/01
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Monogenic Obesity; Non Syndromic Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient cohort: Patients already tested for monogenic obesity with the 71 genes panel.
- Control cohort: Patients tested for other indication than monogenic obesity in the lab. The DNA samples will be sequenced for the 71 obesity genes especially for the study.
  Interventions: Biological: monogenic obesity

INTERVENTIONS:
Biological: monogenic obesity — The DNA samples will be sequenced for the 71 obesity genes especially for the study.
  Groups: Control cohort

SUMMARY:
Non-syndromic monogenic obesity is a group of rare diseases characterized by severe and early onset obesity. Genetic characterization of these rare forms is important to target patients who may benefit from a personnalized care (new treatments, prognosis, adapted hygienic and dietary rules). This study aims to expand the diagnostic analysis from five to 71 genes and additionnaly to refine the causal role of some genes not widely tested in routine practice.

DETAILED DESCRIPTION:
Obesity is a frequent disease mainly caused by environmental/polygenic factors and more rarely caused by the alteration of a single gene ("monogenic obesity"). The diagnosis of these rare forms can lead to personalized management (new treatments, prognosis, adapted hygienic and dietary rules) and family screening. The genetic analysis of monogenic obesity classically includes the five best known genes of the leptin-melanocortin pathway: LEP, LEPR, POMC, PCSK1 and MC4R. The limitation to these five genes allows the diagnosis of only 1 to 3% of monogenic obesity. The use of a genetic panel covering more known causes of monogenic obesity on a pediatric cohort of severe and early obesity will allow to evaluate the relevance of enlarged analyses to adapt the management of these rare diseases. In addition, the penetrance and mode of transmission of some genes related to monogenic obesity remain to be precised.

The study aims to analyze the sequencing of 71 genes related to monogenic obesity in a cohort of 100 patients with early (<6 years) and severe obesity. The clinical and biological phenotype of each case will be documented by retrospective medical datas. Concurrent analysis of a cohort of 100 patients with normal BMI (" control ") aims to better define the genes and transmission patterns with significant penetrance in obesity.

The study will include a first part aiming at including patients and controls in the study for which the Biochemistry laboratory of the Bordeaux University Hospital already has a DNA sample (maximum duration 24 months). The patient cohort will be composed of cases that have already benefited from the genetic analysis of the panel of 71 genes as part of their care. The control cohort will be sequenced for the study. The list of 71 genes comes from the recommendations of the French National Plan of Care regarding obesity of rare causes, adding the genes involved in Bardet Biedl Syndrome. The second step of the work will be to collect the clinical, biological and genetic datas of the patient and control cohorts. The third step will be the datas analyse.

ELIGIBILITY:
o For Patient cohort :

Inclusion criteria:

* Body mass index above the International Obesity Task Force 30 curve by age 6.
* Consent for genetic testing signed with agreement to use secondary data for research purposes.

Exclusion criteria : Opposition of the patient to the research - This opposition of the patient must be received by the investigator of the center within a maximum of 1 month after the sending of the information note.

o For Control cohort :

Inclusion criteria:

* Body mass index under 25 kg/m2 after age 18 and no history of obesity.
* Signed consent for genetic testing with agreement to use biological samples and secondary data for research purposes.

Exclusion criteria:

* Opposition of the patient to the research - This opposition of the patient must be received by the investigator of the center within a maximum of 1 month after the sending of the information note.
* Degraded DNA

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Patient cohort : Patients already tested for monogenic obesity with the 71 genes panel.
  * Control cohort : Patients tested for other indication than monogenic obesity in the lab. The DNA samples will be sequenced for the 71 obesity genes especially for the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Positive rate of patients diagnosed with definite monogenic obesity | inclusion visit
  Positive rate of patients diagnosed with definite monogenic obesity by genetic analysis with the 71 genes panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No